CLINICAL TRIAL: NCT02045901
Title: A Multicenter Trial of the Efficacy and Safety of Diclegis® for Nausea and Vomiting of Pregnancy in Pregnant Adolescents
Acronym: PED-301
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Duchesnay Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PED-301
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Morning Sickness
Keywords: Nausea; Vomiting; Pregnancy; Adolescent; Diclegis; Morning; Sickness
MeSH Terms: conditions — Morning Sickness; Nausea; Vomiting | interventions — dicyclomine, doxylamine, pyridoxine drug combination; Exercise; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclegis (Active Comparator): Participants will be randomized to receive Diclegis or placebo. On Day 1, all participants will take 2 tablets of study drug at bedtime. On Days 2 to 14, participants will take 2 tablets of study drug at bedtime. The minimum dosage will be 2 tablets daily at bedtime, increasing, when indicated, to the maximal dosage of 4 tablets per day on Days 3 to 14.
  Interventions: Drug: Diclegis
- Placebo (Placebo Comparator): Participants will be randomized to receive Diclegis or placebo. On Day 1, all participants will take 2 tablets of study drug at bedtime. On Days 2 to 14, participants will take 2 tablets of study drug at bedtime. The minimum dosage will be 2 tablets daily at bedtime, increasing, when indicated, to the maximal dosage of 4 tablets per day on Days 3 to 14.
  Interventions: Drug: Placebo (Sugar Pill)

INTERVENTIONS:
Drug: Diclegis — On Day 1, all participants will take 2 tablets of Diclegis at bedtime. On Days 2 to 14, participants will take 2 tablets of Diclegis at bedtime. The minimum dosage will be 2 tablets daily at bedtime, increasing, when indicated, to the maximal dosage of 4 tablets per day on Days 3 to 14.
  Other Names: Active
  Arms: Diclegis
Drug: Placebo (Sugar Pill) — On Day 1, all participants will take 2 tablets of Placebo at bedtime. On Days 2 to 14, participants will take 2 tablets of Placebo at bedtime. The minimum dosage will be 2 tablets daily at bedtime, increasing, when indicated, to the maximal dosage of 4 tablets per day on Days 3 to 14.
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the efficacy of Diclegis for the treatment of nausea and vomiting of pregnancy (NVP) in pregnant adolescents aged 12 to 17 years with placebo.

The secondary objective of this study is to compare the safety of Diclegis in pregnant adolescents aged 12 to 17 years with placebo by assessing differences in the severity and occurrence of maternal adverse events (AEs).

DETAILED DESCRIPTION:
This is a multicenter study in the treatment of NVP that will actively recruit pregnant adolescents from approximately 14-16 study sites in the United States. After obtaining informed consent on Day 1, a medical examination will be conducted to ensure eligibility. Participants will be randomized to receive Diclegis or placebo. On Day 1, all participants will take 2 tablets of study drug at bedtime. On Days 2 to 14, participants will take 2 tablets of study drug at bedtime. The minimum dosage will be 2 tablets daily at bedtime, increasing, when indicated, to the maximal dosage of 4 tablets per day on Days 3 to 14. Participants will be required to complete a diary daily to assess the severity of their NVP by using the validated Pregnancy Unique Quantification of Emesis (PUQE) and to record any AEs experienced; the Global Assessment of Well being scale will be completed only on Days 1, 8 and 15. Participants will receive telephone calls daily to assess whether the current dosing regimen is sufficient at relieving NVP symptoms, to review study procedures, and to address her questions/concerns. Participants will return to the clinic for evaluation on Day 4 (±1 day) and Day 15 (±1 day) for an end of study visit.

Eligible participants are those between 12 and 17 years of age, pregnant with a gestational age of 7 to 15 weeks + 0 days, suffering from NVP, with a PUQE score ≥6, and who have not responded to conservative management consisting of dietary/lifestyle advice according to the 2004 American College of Obstetrics and Gynecology (ACOG) Practice Bulletin.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a pregnant female between the following ages: at least 12 years on the day of recruitment (ie, Day 1) and not yet 18 years on the last day of the study (ie, Day 15).
2. The participant must provide written informed consent and/or assent to participate in the study, and agrees that she will follow dosing instructions and complete all required study visits.
3. The participant's entry ultrasound indicates a viable pregnancy and confirms gestational age of the fetus is 7-15 weeks + 0 days at the anticipated time of the first dose of study drug provided that her NVP symptoms began </= 10 weeks gestation. If an ultrasound was performed within 4 weeks of the study entry visit, and results can be obtained, an additional ultrasound is not necessary.
4. The participant is suffering from NVP and has a PUQE score ≥6.
5. The participant has not responded to conservative management consisting of dietary/lifestyle advice according to the 2004 ACOG Practice Bulletin.
6. The participant agrees, if on a multivitamin, to continue on her current dose of multivitamin for the duration of the trial.
7. The participant does not plan termination of the pregnancy.
8. On the basis of medical history, physical examination and screening laboratory tests, the participant is judged to be in good health.
9. The participant must be able to swallow the study drug whole (ie, without splitting, crushing, or chewing the tablets).

Exclusion Criteria:

1. The investigator confirms the participant's nausea and vomiting is of etiology other than NVP.
2. The participant has gestational trophoblastic disease or multifetal gestation.
3. The participant has a condition for which antihistamines, in the opinion of the investigator, are contraindicated (eg, epilepsy, alcoholism, glaucoma, chronic lung disease, urinary retention, and heart block).
4. The participant has a known hypersensitivity to doxylamine succinate other ethanolamine derivative antihistamines, pyridoxine hydrochloride, or any inactive ingredient in the Diclegis or placebo formulation.
5. The participant is taking a monoamine oxidase inhibitor.
6. The participant has used antihistamines, anticholinergics, dopamine antagonists, serotonin antagonists, ginger, or anti-emetic therapy (including acupressure, acupuncture, homeopathic remedies, medical hypnosis, and relief bands) to treat NVP in the previous 48 hours or plans to do so during the study.
7. The participant is using drugs that have anticholinergic activity (eg, tricyclic antidepressants).
8. The participant is taking multivitamins containing more than 10 mg of vitamin B6 or plans to do so during the study.
9. The participant is taking supplementary vitamin B6 in addition to any multivitamin preparation or plans to do so during the study (e.g, total vitamin B6 greater than 10 mg).
10. The participant is currently drinking any amount of alcohol.
11. The participant has any condition that might interfere with the conduct of the study, in the opinion of the investigator. For example, Diclegis® should be used with caution in females with asthma, increased intraocular pressure, narrow angle glaucoma, stenosing peptic ulcer, pyloroduodenal obstruction and urinary bladder-neck obstruction.
12. The participant is likely to be unable to comply with study procedures because of inadequate cognitive or language skills.
13. The participant has received an investigational drug within 30 days before enrollment in this study or is scheduled to receive an investigational drug during the course of this study.
14. The participant is currently breastfeeding.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Nausea and Vomiting of Pregnancy Severity from Baseline to Day 15 | Day 1-Day 15
  The primary objective of this study is to compare the efficacy of Diclegis for the treatment of nausea and vomiting of pregnancy (NVP) in pregnant adolescents aged 12 to 17 years with placebo. NVP severity will be compared using the change in PUQE and Global Assessment of Well-being scores from baseline (Day 1) to Day 15 between adolescents randomized to Diclegis and placebo for 14 days.

SECONDARY OUTCOMES:
Severity and occurences of maternal adverse events | Day 1-Day 15
  The secondary objective of this study is to compare the safety of Diclegis in pregnant adolescents aged 12 to 17 years with placebo by assessing differences in the severity and occurrence of maternal adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — Hospital for Sick Children, 555 University Avenue, Toronto ON Canada, M5G-1X8; Gary Hankins, MD, Principal Investigator — University of Texas Medical Branch, Obstetrics/Gynecology, Route 0587, Galveston Texas USA, 77550-0587
Locations (8):
- United States (8):
  - Watching Over Mothers and Babies, Tucson, Arizona
  - Clinica Del Socorro Medical Group, Inc., Los Angeles, California
  - Futura Research, Norwalk, California
  - Medical Professional CR Center, Miami, Florida
  - Empire Clinical Research, LLC, Miami Lakes, Florida
  - Western Michigan University Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Complete Healthcare for Women, Columbus, Ohio